CLINICAL TRIAL: NCT07188818
Title: A Post-market-clinical Follow-up Investigation of Safety and Performance of Decoria® Essence
Brief Title: Clinical Investigation on Lips Treated With HA-filler
Acronym: DAG-ESS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bohus Biotech AB (Industry)
Collaborators: Key2Compliance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIV-24-04-046794
Record Dates: First submitted 2024-12-19; First posted 2025-09-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Aesthetic Correction of the Lips
Keywords: lips profile; lip augmentation; correction of perioral rhytids; lip volume; lip contour

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational Medical Device (Other): All eligible subjects desiring improvement and correction of their lip profile will receive injection of Decoria Essence in either one or both lips (upper, lower) and/or vermillion lines and/or perioral wrinkles/rhytids.
  Interventions: Device: Decoria Essence

INTERVENTIONS:
Device: Decoria Essence — Decoria® Essence is a hyaluronic acid based, BDDE-crosslinked dermal filler. Decoria® Essence dermal fillers are injected into dermal tissue to improve the volume and the contouring of the lips to desired level of correction by supporting the overlying tissue. Injection volume will be determined by the treating investigator according to the instructions for Use (IFU).

SUMMARY:
A post-market-clinical follow-up investigation to confirm the clinical safety and performance profile of Decoria® Essence for the correction and improvement of lips profile.

DETAILED DESCRIPTION:
A post-market, open-label, prospective, interventional, confirmatory, evaluator-blinded, multi - centre, clinical investigation to confirm the clinical safety and performance profile of Decoria® Essence for the correction and improvement of lips profile.

Subjects desiring correction and improvement of their lip profile at the participating sites will be asked to participate in the clinical investigation. According to national legislation, all subjects must have a consultation with the respective clinic and receive both oral and written information at least 48 hours prior to treatment with fillers, as to allow for sufficient reflection time.

If the subject decides to participate, the subject will receive treatment on Day 0 (Visit 1). At 1 month visit (Visit 2) an optional touch-up may be given as well as assessments performed. All subjects will be followed for 6 months with follow-up and assessments by visits in the clinic (Visit 2, Visit 3 and Visit 4).

Standardized facial photography will be taken prior to and after treatment during Visit 1 and 2 and during each follow-up visit at the clinic (Visit 3, Visit 4 and Visit 5). The photographs will be used for the evaluation of the primary efficacy endpoint of the blinded-evaluator using the Global Aesthetic Improvement Scale (GAIS) as well as the exploratory instrumental evaluation of the lip contour. GAIS will be used for blinded-evaluator assessment, treating Investigator assessment and patient satisfaction.

Numeric Pain Rating Scale (NRS) at each visit involving an injection (Visit 1 and Visit 2 - optional touch up) will be used to measure pain.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years, males and females.
2. Able and willing to give written informed consent for participation in the investigation.
3. Treating investigator considers the subject's lips amenable to an improvement of at least 1 grade on the GAIS. At least one lip should either have a potential to change (augmentation, contouring or both) or have moderate to severe volume deficit. The grades do not have to be the same on both lips.
4. Ability to follow study instructions and likely to complete all required visits.

Exclusion Criteria:

1. Pregnant or lactating females.
2. Any previous hypersensitivity reaction to any constituent of the Investigational medical device (IMD) or to local anaesthetic products.
3. Performed or planned surgery below the nose, permanent implant, injection with fat, and deoxycholic acid that may confound the evaluation of safety and performance of the IMD.
4. Any other intradermal injection, such as semi-permanent fillers or botulinum toxins (no complications are allowed), received in the same injection area within 9 months of the Treatment visit (Visit 1) that may confound the evaluation of safety and performance of the IMD.
5. Has an ongoing episode/relapse, recently diagnosed or newly started medication of an autoimmune disease, as judged by the investigator.
6. Has any chronic or acute skin disease or inflammation (such as pimples, rashes, or hives) within or close to the treatment area.
7. Has any treatments (thrombolytics, anticoagulants etc) or disease related to the coagulation system.
8. Subjects that have taken any type of vaccine within two weeks prior injection with the IMD.
9. Subjects receiving interferon and ribavirin treatment.
10. Features that may interfere with the visual assessment such as recent cosmetic treatment, scarring, abscess, piercing or tattoo below the nose.
11. Participation in a clinical investigation that may affect the safety or performance of this investigation, as judged by the Principal Investigator, or authorized designee.
12. Employees of the study site or the sponsor directly involved with the conduct of the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Primary efficacy endpoint to measure the change/improvement in score using the Global Aesthetic Improvement Scale (GAIS) | From pre-intervention baseline (Visit 1, Day 0) to month 3 (Visit 3, Day 90).
  The primary efficacy endpoint is to measure the change/improvement in score from pre-treatment baseline to 3 months post treatment by an independent evaluator, using the Global Aesthetic Improvement Scale (GAIS). GAIS is a comparative scale, based on assessment of change since before pre-intervention, ranges from 1 (exceptional improvement) to 4 (unaltered) and 5 (worse). The blinded evaluator will compare the pre-intervention face to post-intervention face and assign the level of improvement in the lips according to the GAIS grading. Each lip (upper and lower) will be assessed independently.
Primary safety endpoint by evaluating Adverse Events | From inclusion until the end of the study (6 months)
  The primary safety endpoint is to assess the safety of Decoria® Essence, evaluated by the incidence, intensity, duration, and time of onset of related adverse events (AEs), including injection site reactions, collected during study duration.

SECONDARY OUTCOMES:
Secondary endpoint evaluating pain by Numeric Pain Rating Scale (NRS) | At baseline (Visit 1, Day 0) and optional touch-up (Visit 2, Day 30)
  Pain will be measured by numerical scale Numeric Pain Rating Scale (NRS) (11-point verbal score completed for each target region treated) for each visit involving an injection. 0 representing "no pain" and 10 indicating the "worst pain imaginable"
Secondary endpoint evaluated improvement by GAIS score | At Visit 1 (Day 0), Visit 2 (Day 30), Visit 3 (Day 90) and Visit 4 (Day 180)
  GAIS (Global Aesthetic Improvement Scale) score at 1- months, 3 months and 6 months post-treatment, as assessed by the treating investigator and blinded evaluator. Scoring from 1-5 equals "very much improved," "much improved," "improved," "unchanged," and "worsened,"
Secondary endpoint by evaluating improvement by GAIS | At Visit 1 (Day 0), Visit 2 (Day 30), Visit 3 (Day 90) and Visit 4 (Day 180)
  GAIS (Global Aesthetic Improvement Scale) score at 1- month, 3- months and 6 months post-treatment, as assessed by the subject. Scoring from 1-5 equals "very much improved," "much improved," "improved," "unchanged," and "worsened,"
Secondary endpoint evaluating treatment related Adverse Events | 30 days after injection of initial treatment (Day 0-30) and optional touch-up (Day 30-60)
  Treatment related adverse events and injection site reactions reported after touch-up should be similar to those reported after initial treatment.
Secondary endpoint by instrumental evaluation of lips by image analysis. | From pre-intervention baseline, to post-treatment at Day 1, 30, 90 and 180 respectively
  Change in lip compared to baseline will be measured after treatment, as well as at 1-month, 3-months and 6 months post-treatment visits. Instrumental evaluation of lips will be done by image analysis. A descriptive analysis of the semi.quantative change from baseline and after treatment will be done. Exploration of correction with other endpoints or measurements such as GAIS will be performed posthoc.
Secondary endpoint evaluated outcome by GAIS score | At Visit 1 (Day 0), Visit 2 (Day 30), Visit 3 (Day 90) and Visit 4 (Day 180)
  GAIS (Global Aesthetic Improvement Scale) score at 1- months, 3 months and 6 months post-treatment, as assessed by the treating investigator and blinded evaluator. Scoring from 1-5 equals "very much improved," "much improved," "improved," "unchanged," and "worsened,"

CONTACTS AND LOCATIONS:
Overall Officials: Lucian Grema, M.D., Principal Investigator — Diagnostiskt Centrum Hud, Konsult LBG vard AB
Locations (6):
- Sweden (6):
  - Advanced Clinic, Gothenburg
  - Svenska Hudkliniker Karlstad, Karlstad
  - Hansa Estetik, Malmo
  - Svenska Hudkliniker, Stockholm
  - Dr Filip, Stockholm
  - Peri Estetik, Västerås